CLINICAL TRIAL: NCT00650728
Title: Esophagus Imaging for Radiofrequency Ablation of Atrial Fibrillation: Comparison of Two Methods
Brief Title: Esophagus Imaging for Radiofrequency Ablation of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Prof. Paul Erne, Luzerner Kantonsspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Esophagus imaging
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Atrial Fibrillation
Keywords: radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: placing gastric tube

SUMMARY:
As the left atrium is in close vicinity to the esophagus, radiofrequency ablation in the left atrium may damage the esophagus and create esophageal perforations and esophageal left atrial fistula. The aim of the present study is to compare different methods for visualization of the esophagus to prevent this complication.

DETAILED DESCRIPTION:
Percutaneous catheter ablation with circumferential pulmonary vein isolation using radiofrequency energy has become an important therapeutic option to treat atrial fibrillation over the last years. Importing images from pre-acquired 3-D CT or MRI scans into the 3-D mapping system with superimposition of the electro-anatomical map is increasingly used. Despite these advances, the interventional electrophysiologist must be aware of potential complications that are associated with this procedure. As the left atrium is in close vicinity to the esophagus, radiofrequency ablation in the left atrium may damage the esophagus and create esophageal perforations and esophageal left atrial fistula. To prevent this lethal complication integration of an esophagus tag into the electroanatomic left atrium map visualizing the anatomic relationship has been studied und reported. Another possibility of visualization of the esophagus is to perform the CT after placing a conventional radio-opaque gastric tube, which provides information about the course of the esophagus in relation to the LA and may be scanned by CT . It has been shown that under normal conditions, if no barium is administered, there is little change in the anatomical relationship between the posterior left atrium and the esophagus during the entire cardiac cycle. However it is not clear whether the position of the esophagus in relation to the left atrium is changing over days.

The aim of the present study is to evaluate whether visualization of the esophagus by placing a conventional gastric tube before performing the CT scan and visualization and integration of the esophagus into the 3-D electro-anatomical map the day before ablation is accurate compared with integration of an esophagus tag into the electroanatomic left atrium map visualizing the anatomic relationship during the radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation undergoing radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of localization of the esophagus in relation to the left atrium | one year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, Study Chair — Luzerner Kantonsspital
Locations (1):
- Kantonsspital Luzern, Department of Cardiology, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Kobza R, Schoenenberger AW, Erne P. Esophagus imaging for catheter ablation of atrial fibrillation: comparison of two methods with showing of esophageal movement. J Interv Card Electrophysiol. 2009 Dec;26(3):159-64. doi: 10.1007/s10840-009-9434-3. Epub 2009 Sep 10. PMID 19757002